CLINICAL TRIAL: NCT06388447
Title: Reconstruction of Deficient Interdental Papilla Using Allogenic Umbilical Cord-Mesenchymal Stem Cells vs. Physiological Saline: A Randomised Controlled Trial
Brief Title: Reconstruction of Deficient Interdental Papilla Using Stem Cells vs Physiological Saline
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCMSC1
Record Dates: First submitted 2023-11-30; First posted 2024-04-29 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Umbilical cord-mesenchymal stem cells (Experimental): Injection of the UC-MSC into the interdental papilla using a standardised 1mL syringe will be done. 0.1mL (2millions cells) will be administered per black triangle. If there are three black triangles, only two black triangle will be treated, skipping the middle black triangle to avoid additive effect of the intervention
  Interventions: Biological: Umbilical cord-mesenchymal stem cells
- Physiological saline (Placebo Comparator): Injection of the 0.9% Sodium chloride (NaCl) into the interdental papilla using a standardised 1mL syringe will be done. 0.1mL of 0.9% NaCl will be administered per black triangle. If there are three black triangles, only two black triangle will be treated, skipping the middle black triangle to avoid additive effect of the intervention
  Interventions: Biological: Umbilical cord-mesenchymal stem cells

INTERVENTIONS:
Biological: Umbilical cord-mesenchymal stem cells — One injection will be given at each papilla set with the volume of 0.1mL with 2.0 x 10⁶ cells per syringe at every visit. A total of 3 injections will be given at the interval of 6 weeks, with a total of 6.0 x 10⁶ cells for each interdental papilla at the end of the 3 injections. Every injection starts with locally application of local anesthetic. For the control group, participants will be injected with 0.9% sodium chloride after locally application of local anesthetic

SUMMARY:
The goal of this study is to assess the reconstruction of interdental papilla following the injection of UC-MSCs or physiological saline in patients with interdental papilla deficiency. Participants will be randomised into 2 groups (intervention vs placebo) to receive the treatment.

DETAILED DESCRIPTION:
This is a two-arm parallel, prospective, single-center randomised clinical trial, which will be designed based on the guidelines from the Consolidated Standards of Reporting Trials (CONSORT) statement and will be registered in clinicaltrials.gov. Participants will be screened according to the inclusion and exclusion study criteria, and recruited from Orthodontic Postgraduate Clinic, Universiti Malaya.

Total sample size will be set at 20 interdental papilla after considering all the sample sizes calculated using different objectives, due to the cost effectiveness, the practicability, and consideration on the risk and complications.

This research is divided into 3 phases: pre-operative, operative, and post-operative phase.

Pre-operative includes full mouth scaling, baseline data collection (intra-oral scanning for soft tissue; cone beam computed tomography (CBCT) for hard tissue, basic periodontal examination). Then, the black triangle from upper or lower arch will be randomly assigned to two groups: the intervention (Stem cells) group, and the control (saline) group.

Operative phase involves injection either with the experimental or control solution. One injection will be given at each papilla set with the volume of 0.1mL with 2.0 x 10⁶ cells per syringe at every visit. A total of 3 injections will be given at the interval of 6 weeks, with a total of 6.0 x 10⁶ cells for each interdental papilla at the end of the 3 injections. Every injection starts with locally application of local anesthetic. For the control group, participants will be injected with 0.9% sodium chloride after locally application of local anesthetic.

Post-operatively, at 6, 12, 24 and 36 weeks, data will be collected for analysis. Intra-oral scanning of soft tissue will be done at every visits. CBCT for hard tissue will be done at 36 weeks. At every follow up, basic periodontal examination will be scored for periodontal health supervision. Data collected will be entered and analysed using SPSS 26.0. Images from the scans (soft tissue scans, hard tissue scans) will be superimposed and the difference between the 2 images will be calculated and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 - 40 years
* Non-smoker
* Able to understand English
* Subjects who are able to attend follow up during the clinical trial
* Subjects who are able to maintain oral hygiene (< 10% FMPS) with BPE score 0, 1, or 2 at the upper anterior or lower anterior sextant
* Subjects having at least one deficient interdental papilla in the upper or lower arch or both in the anterior region (from canine to contralateral canine) with papillary deficiency type I or II, according to Nordland and Tarnow classification
* No history of regular medication intake (nifedipine, calcium channel blockers, cyclosporine, phenytoin, etc)
* Teeth free from caries, proximal restorations, fixed prosthesis or orthodontic fixed appliances (except for fixed retainer that does not encroach on black triangle)
* No open contacts between affected teeth
* No history of periodontal surgical or non-surgical treatment (Root surface debridement) over the last six months at the area of interest
* Probing pocket depth ≤ 4mm without bleeding on probing at the area of interest

Exclusion Criteria:

* Passive smoker/ former smoker/ electronic smoker
* Alcoholic
* Pregnant or breastfeeding females
* Subjects with current or previous drug intake that may predispose to gingival enlargement (nifedipine, calcium channel blockers, cyclosporin, phenytoin, etc)
* Subjects with medical conditions that may affect periodontal healing/ Reconstruction (diabetes, cardiovascular disease, stroke, asthma)
* Subjects with physical impairment, orofacial deformities
* Subjects with documented drug allergic, or history of allergic reaction to any constituents of injection
* Subjects who had active or past history of neoplasia
* Subjects who are on active orthodontic treatment/ require active tooth movement at the area of interest
* Subjects with probing pocket depth of more than 4mm with bleeding on probing at the area of interest
* Subjects with full mouth plaque score >10%
* Subjects with a history of periodontal surgical or non-surgical treatment over the last six months at the area of interest

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Volumetric difference of the deficient interdental papilla pre- and post-intervention | 9 months
  Intra-oral scanner will be used to scan the dentition and gingiva. Both pre- and post- intervention scans will be exported to Materialise 3-matics software to be superimposed and analyse for the volumetric difference
Volumetric difference of the interdental bone between pre- and post-intervention | 9 months
  Cone beam computed tomography (CBCT) will be taken before intervention and 9 months after intervention. The CBCT images will be exported to Materialise 3-matics software to be superimposed and volumetric difference would be analysed.
Difference of bone density between pre-and post- intervention | 9 months
  CBCT will be taken pre-intervention and 9 months after intervention. The CBCT images will be exported to Materialise 3-matics software. A range of "hu" will be selected as "old bone". Different in bone density from the range indicates new bone formation.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthodontic Postgraduate Clinic, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No